CLINICAL TRIAL: NCT00429585
Title: Intramedullary Nail Versus Plate Fixation Re-Evaluation Study in Proximal Tibial Fractures: A Multicenter Randomized Trial Comparing IM Nails and Plate Fixation (IMPRESS)
Brief Title: A Multicenter Randomized Trial Comparing IM Nails and Plate Fixation in Proximal Tibial Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Orthopaedic Trauma Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-25923
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Results first posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Tibial Fractures
Keywords: tibia fracture; proximal tibia; interlocking intramedullary nail; locking periarticular plate; open reduction; internal fixation
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Randomized Treatment - Nail (Other): Randomized Treatment - Nail
  Interventions: Device: reamed, interlocking intramedullary nail
- Randomized Treatment - Plate (Other): Randomized Treatment - Plate
  Interventions: Device: locking periarticular plate

INTERVENTIONS:
Device: reamed, interlocking intramedullary nail — Standard of care device for tibia fracture repair; Randomized Treatment - Nail
  Arms: Randomized Treatment - Nail
Device: locking periarticular plate — Standard of care device for tibia fracture repair; Randomized Treatment - Plate
  Arms: Randomized Treatment - Plate

SUMMARY:
This study looks at two types of surgical treatments and hopes to answer the question: which is the best way to surgically treat a proximal tibia fracture? Both procedures being studied are standard of care (used routinely) and use FDA approved devices. All medical and surgical treatment will be the same for participants as non-participants.

DETAILED DESCRIPTION:
The study is a multicenter randomized controlled trial in which individuals sustaining a fracture of the proximal metaphysis of the tibia will be operatively managed by one of two strategies. The first strategy involves fixation of the fracture with a reamed, interlocking intramedullary nail (Nail Group). The second treatment strategy involves open reduction and internal fixation of the fracture with a locking periarticular plate (Plate Group). The null hypothesis of the study is that there will be no difference in the two groups with respect to the primary and secondary outcome measures. To the degree possible, patients in the two groups will receive post-operative care according to the same standards and protocols.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature,
* Extra-articular fracture of the proximal tibia extending into the metaphyseal with or without intra-articular extension not requiring open reduction with complete anteroposterior (AP) and lateral radiographs,
* Major fracture line not closer than 4cm from the proximal tibial articular surface
* Fracture requiring operative treatment amenable to either IM nail or plate
* Surgeon agreed to randomize patient
* Informed consent obtained
* Patient is English speaking

Exclusion Criteria:

* Tibial shaft fractures not amenable to intramedullary nailing (i.e.fracture is less than 4 cm from joint surface),
* Fracture of the proximal tibia with intraarticular extension requiring open reduction,
* Known metabolic bone disease
* Separate displaced tibial tubercle fragment,
* Soft tissue injuries compromising treatment method with nail,plate or both.
* Fractures with vascular injury (Gustillo Type IIIC injury) requiring repair,
* Compartment syndrome of the leg diagnosed preoperatively,
* Pathological fractures,
* Retained hardware or existing deformity in the affected limb that would complicate IM nailing,plating or both,
* Symptomatic knee arthritis.
* Surgical delay greater than 3 weeks for closed fractures or 24 hours for open fractures,
* Immunocompromised,
* Unable to comply with postoperative rehabilitation protocols or instructions (i.e. head injured or mentally impaired),
* Current or impending incarceration,
* Unlikely to follow-up in surgeon's estimation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2007-02 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Tornetta, M.D., Principal Investigator — Boston University
Locations (29):
- United States (27):
  - University of Alabama - Burmingham, Birmingham, Alabama
  - University of California at Davis, Davis, California
  - University of California-San Francisco, San Francisco, California
  - Tampa General Hospital, Tampa, Florida
  - Indiana University, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Orthopaedic Associates of Michigan, Grand Rapids, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - St. Mary's Hospital - Mayo Clinic, Rochester, Minnesota
  - Barnes Hospital, St Louis, Missouri
  - St. Louis University Hospital, St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - New York Hospital for Joint Diseases, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Oklahoma/ Health Science, Oklahoma City, Oklahoma
  - Oregon health and science university, Portland, Oregon
  - University Of Pittsburgh, Pittsburgh, Pennsylvania
  - Campbell Foundation, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Orthopaedic Specialty Associates - Fort Worth, Fort Worth, Texas
  - Harborview Medical Center, Seattle, Washington
- Canada (2):
  - Victoria Hospital, London, Ontario
  - St. Michaels Hospital - Toronto, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 9 participants were enrolled but were not randomized. Of those 9, 6 were found ineligible after consent and 3 withdrew consent prior to randomization.
Period: Overall Study
Arm/Group | Randomized Treatment - Nail | Randomized Treatment - Plate
Started | 52 | 47
Completed | 22 | 27
Not Completed | 30 | 20
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 27 | 20
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized Treatment - Nail | Randomized Treatment - Plate | Total
Number analyzed (Participants) | 52 | 47 | 99
Age, Continuous [Mean (Full Range); unit: years] | 43 [20 to 74] | 48 [20 to 87] | 46 [20 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 40 | 36 | 76
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 52 | 47 | 99

OUTCOME MEASURES:

1. Primary Outcome: Participants' Quality of Life at 3 Months
Description: The European Quality of Life Five Dimension (EQ-5D) Survey will be used to measure the participants' quality of life. The EQ-5D measures the subjects' overall state, including 5 domains: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3=moderate problems, 4=severe problems and 5=extreme problems. The score is determined by a scale and grading systems that can range from 0.01 to 1.00. The lower the score the less quality of life problems.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Treatment - Nail | Randomized Treatment - Plate
Number analyzed (Participants) | 46 | 38
score on a scale | 0.60 (0.24) | 0.59 (0.20)

2. Primary Outcome: Participants' Quality of Life at 6 Months
Description: as for outcome 1
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Treatment - Nail | Randomized Treatment - Plate
Number analyzed (Participants) | 43 | 38
score on a scale | 0.65 (0.19) | 0.72 (0.20)

3. Primary Outcome: Participants' Quality of Life at 12 Months
Description: The European Quality of Life Five Dimension (EQ-5D) Survey will be used to measure the participants' quality of life. The EQ-5D measures the subjects' overall state, including 5 domains: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3=moderate problems, 4=severe problems and 5=extreme problems. The score is determined by a scale and grading systems that can range from 0.01 to 1.00. The higher the score the less quality of life problems.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Treatment - Nail | Randomized Treatment - Plate
Number analyzed (Participants) | 22 | 27
score on a scale | 0.60 (.24) | 0.775 (0.16)

4. Primary Outcome: Injury Related Limitations and Concerns at 3 Months
Description: Participant limitations and bother from the injury will be assessed using the Short Musculoskeletal Function Assessment (SMFA).This survey asks the subject 46 questions, they are broken up into 2 parts. Part 1 relates to the difficulty/limitations the subject has related to their injury. Part 2 is how much the subject is bothered by this injury. Subjects provide score on a scale of 1 (no difficulty/bother) to 5 (highly difficult/bothered). The scoring range is between 0-100. The lower the score the less injury related limitations and bother.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Treatment - Nail | Randomized Treatment - Plate
Number analyzed (Participants) | 46 | 38
score on a scale | 40.25 (19.74) | 40.11 (16.28)

5. Primary Outcome: Injury Related Limitations and Concerns at 6 Months
Description: as for outcome 4
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Treatment - Nail | Randomized Treatment - Plate
Number analyzed (Participants) | 43 | 38
score on a scale | 32.19 (18.70) | 27.70 (18.58)

6. Primary Outcome: Injury Related Limitations and Concerns at 12 Months
Description: Participant limitations and bother from the injury will be assessed using the Short Musculoskeletal Function Assessment (SMFA).This survey asks the subject 46 questions, they are broken up into 2 parts. Part 1 relates to the difficulty/limitations the subject has related to their injury. Part 2 is how much the subject is bothered by this injury. Subjects provide score on a scale of 1 (no difficulty/bother) to 5 (highly difficult/bothered). The scoring range is between 0-100. The lower the score the less difficulty and bother.
Time Frame: 12 month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Treatment - Nail | Randomized Treatment - Plate
Number analyzed (Participants) | 22 | 27
score on a scale | 34.20 (20.93) | 23.51 (19.35)

7. Secondary Outcome: Number of Participants With Fracture Nonunions
Description: A nonunion is when a broken bone fails to heal. This is determined by a review of the participants' medical records and x-rays.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Treatment - Nail | Randomized Treatment - Plate
Number analyzed (Participants) | 22 | 27
Participants | 4 | 5

8. Secondary Outcome: Number of Participants With Superficial Infections
Description: A superficial infection is an infection that occurs at the wound only. Participants are monitored during clinical exams throughout the 12 month follow up appointments and medical records are reviewed.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Treatment - Nail | Randomized Treatment - Plate
Number analyzed (Participants) | 43 | 38
Participants | 0 | 2

9. Secondary Outcome: Number of Participants With Deep Infections
Description: A deep infection is an infection occurring at the site of the nail or plate. Participants are monitored during clinical exams throughout the 12 month follow up appointments and medical records are reviewed.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Treatment - Nail | Randomized Treatment - Plate
Number analyzed (Participants) | 43 | 38
Participants | 3 | 1

10. Secondary Outcome: Number of Participants With Compartment Syndrome
Description: Compartment syndrome is a painful condition that occurs when pressure within the muscles builds to dangerous levels. Participants are monitored during clinical exams throughout the 12 month follow up appointments and medical records are reviewed.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Treatment - Nail | Randomized Treatment - Plate
Number analyzed (Participants) | 43 | 38
Participants | 1 | 0

11. Secondary Outcome: Number of Participants With Malunion (>5 Degrees Varus/Valgus)
Description: Malunion is when a broken bone heals in an abnormal position. In this case, more than a 5 degree angle varus (curving into) or valgus (curving away). This is determined by a review of the participants' medical records and x-rays.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Treatment - Nail | Randomized Treatment - Plate
Number analyzed (Participants) | 22 | 27
Participants | 3 | 3

ADVERSE EVENTS:
Time Frame: 6 years
Description: Adverse event information was collected during clinical followup appointments through questionnaires/surveys.
Arm/Group | Randomized Treatment - Nail | Randomized Treatment - Plate
All-Cause Mortality (participants affected / at risk) | 1/52 | 0/47
Serious Adverse Events (participants affected / at risk) | 4/52 | 2/47
Other Adverse Events (participants affected / at risk) | 16/52 | 13/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Treatment - Nail (N=52) | Randomized Treatment - Plate (N=47)
Patient fall (Surgical and medical procedures) | 1 (1) | 0 (0) — Patient fell post op day 1 with catastrophic failure of proximal fixation requiring revision surgery
Fracture (Surgical and medical procedures) | 1 (1) | 1 (1) — Extraarticular pilon fracture at distal end of nail requiring orif; Non displaced Dist.Fibula Fx
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Over 1 yr since study enrollment. Patient has osteoporosis contralateral distal femur fracture after low energy fall.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — ASPIRATION PNEUMONIA
Death (Cardiac disorders) | 1 (1) | 0 (0) — Multitrauma/Stroke/Intracranial Hypertension
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Treatment - Nail (N=52) | Randomized Treatment - Plate (N=47)
Painful Implant (Surgical and medical procedures) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 3 (3) | 3 (3)
Nonunion (Surgical and medical procedures) | 4 (4) | 5 (5)
Malunion (Surgical and medical procedures) | 3 (3) | 3 (3)
Wound Breakdown Right Proximal Tibia Surgical Site (Surgical and medical procedures) | 2 (2) | 0 (0)
Anterior compartment not functional (Surgical and medical procedures) | 1 (1) | 0 (0)
Delayed Union (Surgical and medical procedures) | 1 (1) | 0 (0) — delayed fracture healing
Peripheral Nerve Injury (Surgical and medical procedures) | 0 (0) | 2 (2)
DVT (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT00429585/Prot_SAP_000.pdf